CLINICAL TRIAL: NCT04353583
Title: Acute Kidney Injury (AKI) and Acute Kidney Disease (AKD) in Patients With Coronavirus Disease 2019 (COVID-19)
Brief Title: Acute Kidney Injury and Acute Kidney Disease in COVID-19
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 58/20
Record Dates: First submitted 2020-04-06; First posted 2020-04-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; Corona Virus Infection
MeSH Terms: conditions — Acute Kidney Injury; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU patients: Inpatients with COVID-19 requiring ICU care
- Non-ICU patients: Inpatients with COVID-19 not requiring ICU care

SUMMARY:
Acute kidney injury (AKI) has been identified as an independent risk factor for in-hospital mortality. The present study aims to investigate the incidence of AKI and renal recovery of inpatients diagnosed with COVID-19.

DETAILED DESCRIPTION:
Beginning in December 2019, a novel coronavirus, designated as severe acute respiratory distress coronavirus 2 (SARS-CoV-2), has caused an international outbreak of respiratory illness termed coronavirus disease 2019 (COVID-19). Although the clinical manifestations of COVID-19 are dominated by respiratory symptoms, some patients show severe kidney abnormalities. Acute kidney injury (AKI) has been identified as an independent risk factor for in-hospital mortality. The present study aims to investigate the incidence of AKI and renal recovery of inpatients diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1) Patients with COVID-19 diagnosed by World Health Organisation (WHO) criteria

Exclusion Criteria:

1. Patients aged less than 18 years
2. Patients with stage 4 chronic kidney disease (baseline estimated glomerular filtration rate <30 ml/min/1.73 m2)
3. Patients receiving maintenance dialysis
4. Recipients of solid-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with diagnosed COVID-19
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI | 30 days post-hospital admission
  Serial assessment of serum creatinine and urine output
Cystatin C as indicator of mortality | 30 days post-hospital admission
  All-cause mortality
Cystatin C as indicator of renal disease | 30 days post-hospital admission
  AKI and acute kidney disease (AKD)
Cystatin C as indicator of respiratory illness | 30 days post-hospital admission
  Ventilator-free days
Cystatin C as indicator of disease severity | 30 days post-hospital admission
  Rate of intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University Hospital Giessen and Marburg, Giessen
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Naicker S, Yang CW, Hwang SJ, Liu BC, Chen JH, Jha V. The Novel Coronavirus 2019 epidemic and kidneys. Kidney Int. 2020 May;97(5):824-828. doi: 10.1016/j.kint.2020.03.001. Epub 2020 Mar 7. No abstract available. PMID 32204907